CLINICAL TRIAL: NCT04292301
Title: Multi-Centered Study Comparison of Output Images From STrategically Acquired Gradient Echo to Conventional 1.5 T and 3.0 T Magnetic Resonance Images and Assessing Their Clinical Usability on Human Participants
Brief Title: MRI Assessing Clinical Usability of STrategically Acquired Gradient Echo on Human Participants
Acronym: STAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SpinTech, Inc. (Other)
Collaborators: Summit Medical Center (Other); Center for Diagnostic Imaging (Other); Loma Linda University (Other); University of Texas Southwestern Medical Center (Other); University of Iowa (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CP-STAGE-001
Record Dates: First submitted 2020-02-25; First posted 2020-03-03 (Actual); Results first posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-05

CONDITIONS: MRI
Keywords: Magnetic Resonance Imaging; Image Post-Processing; Neuro-Radiology

STUDY DESIGN:
Intervention Model Description: All human participants in the study will be imaged using MRI under the same acquisition protocol. The STAGE protocol is collected alongside conventional MR.
Masking Description: Study does not involve masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- STrategically Acquired Gradient Echo (STAGE) (Experimental): STAGE Inputs are flow compensated 3D gradient echo MR images acquired at optimal parameters which are used to calculate multiple contrasts for brain imaging. All subjects within the study are imaged using both a conventional MR protocol and STAGE protocol.
  Interventions: Device: STrategically Acquired Gradient Echo (STAGE)

INTERVENTIONS:
Device: STrategically Acquired Gradient Echo (STAGE) — The STAGE package uses conventional 3D gradient echo MR, its magnitude and phase, collected at set parameters which allow for the reconstruction of multiple MR datasets which results in decreased acquisition time, equivalency to conventional MR, and the decrease in scan time allows for a higher standard of wealth within the data acquired.

SUMMARY:
The study's purpose is to validate STAGE images and, when applicable, their equivalence to conventional MRI through an assessment by a trained certified neuroradiologist in a clinical setting. For STAGE images without conventional equivalent, the neuroradiologist will determine if their contrasts, intensities, and quality are sufficient and meet expectations for images used in radiological reads of the brain. The study is a multi-center study in which STAGE can be assessed at sites with different MRI manufacturers and field strengths. Site names will be made available to the collaborators and participants. The sponsor is based out of Michigan, while participating sites may be located in other states. Any funding for the study will come from an industry source, SpinTech, Inc.

DETAILED DESCRIPTION:
The scope of the study includes the acquisition of MR images from a specified MR manufacturer, the installation of the STAGE device at the clinical site, the subsequent processing of the acquired MR images, and their evaluation by neuroradiologists. The follow section will summarize the key procedures which are involved in this study.

1. Participants will be enrolled as study subjects per IRB approved protocol and informed consent.
2. The STAGE device will be installed at the clinical site. The installation of the Investigational STAGE module requires it to be labeled for Investigational Use Only, per FDA requirements. It requires an available power source and live Ethernet connection. STAGE is connected to the PACS via a node which requires the AE title and an assigned IP address. The node will only accept images which meet the STAGE protocol requirements and any other images are not used. After the images are processed and sent back to the PACS system, all data are purged from the STAGE module. A log is kept of which data was processed which can be viewed through the assigned IP within a web browser. All images under the study protocol shall be labeled "For Investigational Device Use Only".
3. The PI and Co-Investigators will be trained on the use of installed STAGE investigational device. This will include a review of the installation and user manuals written as documentation under the FDA regulated development process. Documentation of the training process will be documented with data workflow and output images being presented.
4. After these steps the clinical study collection of MR images will begin. Since a primary aim of STAGE is to reduce acquisition times while generating a wealth of contrasts from the dataset, additional conventional MR images will be acquired including but not limited to: T1W, Susceptibility Weighted Images (SWI), Magnetic Resonance Angiography (MRA), and Spin Density Weighted (PDW). The patient's time in the magnet will be kept under 40 minutes. The STAGE protocol is available for Siemens, GE, Philips, and Canon/Toshiba magnets at both 1.5T and 3.0T field strengths. The processed STAGE images will be sent back to the PACS system where they remain within the participant's scan folder and are clearly labeled. They can then be viewed at an integrated workstation.
5. The study data will then be collected on Case Report Forms to record the response from the reading radiologist as well as the documented acquisition times for the STAGE protocol and the standard of care acquisition times used within that clinical setting (control arm of study). Prospective data will include imaging as well as questionnaire/survey with the radiologist to evaluate the performance of STAGE and its outputs. The study will not consist of retrospective data.
6. Clinical study completions and closeout. At the conclusion of the study, STAGE will be removed from the site by a trained technician and all data from the study will be purged from the PACS. A checklist will be documented to show that all measurable clinical response metrics have been recorded and that the study has successfully contributed its intended aims while following IRB and FDA regulations for clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 6-80 years of age, inclusive.
* Literate in English
* No contraindications to MR
* Not claustrophobic

Exclusion Criteria:

* Subject has diffuse white matter disease or leukoaraiosis.
* Participant, or if participant is under 18 years of age, participant's parent or guardian unable to read and sign an informed consent.
* Women who are pregnant or breast-feeding.
* Those with major surgery within the past eight weeks or scheduled surgery within 30 days.
* Chronic back pain or inability to lie still for 5 minutes or more.
* History of drug or alcohol abuse.
* Individuals who exceed 28 BMI or 320 lbs.
* Individual whose girth exceeds the magnetic bore.
* Direct employee or student of the PI.
* Participants belong to a vulnerable group.

Ages: 6 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2021-01-07 (Actual); Study Completion 2021-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas P Beall, MD, Principal Investigator — Summit Medical Center; Murray A Solomon, MD, Principal Investigator — Center for Diagnostic Imaging; Vincent Magnotta, MD, Principal Investigator — University of Iowa; Karen Tong, MD, Principal Investigator — Loma Linda University Health; Frank Yu, MD, Principal Investigator — University of Texas; Letterio Politi, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (5):
- United States (5):
  - Loma Linda University Health, Loma Linda, California
  - Insight Imaging - Center for Diagnostic Imaging, Los Gatos, California
  - University of Iowa, Iowa City, Iowa
  - Summit Medical Center, Edmond, Oklahoma
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haacke EM, Chen Y, Utriainen D, Wu B, Wang Y, Xia S, He N, Zhang C, Wang X, Lagana MM, Luo Y, Fatemi A, Liu S, Gharabaghi S, Wu D, Sethi SK, Huang F, Sun T, Qu F, Yadav BK, Ma X, Bai Y, Wang M, Cheng J, Yan F. STrategically Acquired Gradient Echo (STAGE) imaging, part III: Technical advances and clinical applications of a rapid multi-contrast multi-parametric brain imaging method. Magn Reson Imaging. 2020 Jan;65:15-26. doi: 10.1016/j.mri.2019.09.006. Epub 2019 Oct 16. PMID 31629075
- [Background] Wang Y, Chen Y, Wu D, Wang Y, Sethi SK, Yang G, Xie H, Xia S, Haacke EM. STrategically Acquired Gradient Echo (STAGE) imaging, part II: Correcting for RF inhomogeneities in estimating T1 and proton density. Magn Reson Imaging. 2018 Feb;46:140-150. doi: 10.1016/j.mri.2017.10.006. Epub 2017 Oct 20. PMID 29061370
- [Background] Chen Y, Liu S, Wang Y, Kang Y, Haacke EM. STrategically Acquired Gradient Echo (STAGE) imaging, part I: Creating enhanced T1 contrast and standardized susceptibility weighted imaging and quantitative susceptibility mapping. Magn Reson Imaging. 2018 Feb;46:130-139. doi: 10.1016/j.mri.2017.10.005. Epub 2017 Oct 19. PMID 29056394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject recruitment took place across three sites and resulted in a total of 92 participant enrollment with 89 participants remaining after attrition. Recruitment took place between July 2020 and December 2020.
Period: Overall Study
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
Started | 92
Completed | 89
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 92 participants were imaged using STAGE and conventional MR protocols. 89 participants were included in the final analysis after an attrition of 3 participants data due to image artifact due to excessive patient motion or acquisition hardware error.
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
Number analyzed (Participants) | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 89
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 39
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 92

OUTCOME MEASURES:

1. Primary Outcome: Numeric Rating Scale of Clinical Usability Assessment of STAGE Outputs
Description: Reading radiologists responses on the clinical usability of STAGE Outputs based on image quality using a numeric rating scale of 1 to 5 with: 1=unacceptable, 2=poor, 3=acceptable, 4=good, 5=excellent. Scores of 3 or greater are considered clinically usable.
Time Frame: Baseline Only
Population: Scores of 3 or greater are considered clinically acceptable. The count of participants is presented for each score and for each STAGE output series.
Measure: Count of Participants; unit: Participants
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
Number analyzed (Participants) | 89
Participants
  Conventional T1W Input Score=5 | 49
  Conventional T1W Input Score=4 | 40
  Conventional T1W Input Score=3 | 0
  Conventional T1W Input Score<=2 | 0
  Conventional PDW Input Score=5 | 44
  Conventional PDW Input Score=4 | 45
  Conventional PDW Input Score=3 | 0
  Conventional PDW Input Score<=2 | 0
  Conventional MPRAGE Score=5 | 49
  Conventional MPRAGE Score=4 | 40
  Conventional MPRAGE Score=3 | 0
  Conventional MPRAGE Score<=2 | 0
  STAGE T1W Score=5 | 49
  STAGE T1W Score=4 | 39
  STAGE T1W Score=3 | 1
  STAGE T1W Score<=2 | 0
  STAGE PDW Score=5 | 36
  STAGE PDW Score=4 | 50
  STAGE PDW Score=3 | 3
  STAGE PDW Score<=2 | 0
  STAGE T1We Score=5 | 49
  STAGE T1We Score=4 | 37
  STAGE T1We Score=3 | 3
  STAGE T1We Score<=2 | 0
  STAGE T1We Coronal Score=5 | 38
  STAGE T1We Coronal Score=4 | 28
  STAGE T1We Coronal Score=3 | 23
  STAGE T1We Coronal Score<=2 | 0
  STAGE T1We Sagittal Score=5 | 44
  STAGE T1We Sagittal Score=4 | 24
  STAGE T1We Sagittal Score=3 | 21
  STAGE T1We Sagittal Score<=2 | 0
  STAGE T1 MAP Score=5 | 48
  STAGE T1 MAP Score=4 | 40
  STAGE T1 MAP Score=3 | 1
  STAGE T1 MAP Score<=2 | 0
  STAGE PD MAP Score=5 | 48
  STAGE PD MAP Score=4 | 39
  STAGE PD MAP Score=3 | 2
  STAGE PD MAP Score<=2 | 0
  STAGE SWI Score=5 | 1
  STAGE SWI Score=4 | 54
  STAGE SWI Score=3 | 34
  STAGE SWI Score<=2 | 0
  STAGE tSWI Score=5 | 3
  STAGE tSWI Score=4 | 55
  STAGE tSWI Score=3 | 31
  STAGE tSWI Score=2 | 0
  STAGE iSWIM Score=5 | 9
  STAGE iSWIM Score=4 | 58
  STAGE iSWIM Score=3 | 21
  STAGE iSWIM Score<=2 | 1
  STAGE R2* MAP Score=5 | 26
  STAGE R2* MAP Score=4 | 35
  STAGE R2* MAP Score=3 | 27
  STAGE R2* MAP Score<=2 | 1
  STAGE T2* MAP Score=5 | 2
  STAGE T2* MAP Score=4 | 35
  STAGE T2* MAP Score=3 | 51
  STAGE T2* MAP Score<=2 | 1
  STAGE MRA Score=5 | 35
  STAGE MRA Score=4 | 27
  STAGE MRA Score=3 | 27
  STAGE MRA Score<=2 | 0
  STAGE pSWIM Score=5 | 34
  STAGE pSWIM Score=4 | 33
  STAGE pSWIM Score=3 | 22
  STAGE pSWIM Score<=2 | 0
  STAGE mpSWIM Score=5 | 36
  STAGE mpSWIM Score=4 | 31
  STAGE mpSWIM Score=3 | 22
  STAGE mpSWIM Score<=2 | 0
  STAGE DIR Score=5 | 45
  STAGE DIR Score=4 | 21
  STAGE DIR Score=3 | 22
  STAGE DIR Score<=2 | 1

2. Primary Outcome: Review of STAGE Outputs for Artifact and Image Contrast
Description: Reading radiologist and image analyst responses on the clinical usability of STAGE Outputs based on image quality using a yes/no criteria for presence of novel or accentuated imaging artifact. Hardware or participant artifact contributions (i.e. coil sensitivity and motion) were not considered unless noted as increased due to the STAGE method. Each image series was evaluated for the presence of artifact. The total count of the artifacts reported across series evaluated in the study is reported.
Time Frame: Baseline Only
Population: Reported number of observed artifacts within image series are shown as a count.
Measure: Number; unit: Artifact Count
Units Other Than Participants: Image Series
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
Number analyzed (Participants) | 89
Number analyzed (Image Series) | 89
Artifact Count
  Conventional T1MPRAGE | 0
  Conventional T1W | 0
  Conventional PDW | 0
  STAGE T1W | 0
  STAGE PDW | 0
  STAGE T1WE | 0
  STAGE T1MAP | 0
  STAGE PDMAP | 0
  STAGE SWI | 0
  STAGE tSWI | 0
  STAGE iSWIM | 0
  STAGE R2*MAP | 0
  STAGE T2*MAP | 0
  STAGE MRA | 0
  STAGE pSWIM | 0
  STAGE mpSWIM | 0
  STAGE DIR | 0

3. Primary Outcome: Review of STAGE Outputs for Expected Brain Structural Appearance
Description: Reading radiologists responses on the clinical usability of STAGE Outputs based on image appearance of specified brain structures using pass/fail criteria. Expected brain contrast between tissue types will vary depending on the output reviewed (i.e. T1W, PDW, SWI). The behavior of tissue contrasts (i.e. white matter vs gray matter) should also demonstrate standard anatomic contrast (T1W, PDW, SWI) as well quantitative ratio for maps (T2*MAP, R2*MAP, SWIM, T1MAP, PDMAP). For artery/vein appearance, STAGE T1W, T1MAP and PD MAP were not evaluated due to artery/vein not appearing in the image contrasts. For GM/WM/CSF, the MRA, pSWIM and mpSWIM were not evaluated due to the anatomic contrast not appearing in the image contrasts. For calcium/iron appearance, T1WE, T1MAP, PDMAP, MRA, and DIR were not evaluated due to the calcium/iron not appearing in the image contrasts.
Time Frame: Baseline Only
Population: Image series were evaluated for 1) correct artery/vein appearance, 2) calcium/iron appearance, and 3) contrast between gray matter, white matter, and cerebrospinal fluid. Data were evaluated across all STAGE output images based on these structures appearance. The count of image series units is shown as either meeting criteria or not.
Measure: Count of Units; unit: Image Series
Units Other Than Participants: Image Series
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
Number analyzed (Participants) | 89
Number analyzed (Image Series) | 89
Image Series
  Artery and Vein: Conventional T1MPRAGE Criteria Met | 89
  Artery and Vein: Conventional T1MPRAGE Criteria Not Met | 0
  Artery and Vein: Conventional T1W Criteria Met | 89
  Artery and Vein: Conventional T1W Criteria Not Met | 0
  Artery and Vein: Conventional PDW Criteria Met | 89
  Artery and Vein: Conventional PDW Criteria Not Met | 0
  Artery and Vein: STAGE T1W Criteria Met | 89
  Artery and Vein: STAGE T1W Criteria Not Met | 0
  Artery and Vein: STAGE PDW Criteria Met | 89
  Artery and Vein: STAGE PDW Criteria Not Met | 0
  Artery and Vein: STAGE SWI Criteria Met | 89
  Artery and Vein: STAGE SWI Criteria Not Met | 0
  Artery and Vein: STAGE tSWI Criteria Met | 89
  Artery and Vein: STAGE tSWI Criteria Not Met | 0
  Artery and Vein: STAGE iSWIM Criteria Met | 89
  Artery and Vein: STAGE iSWIM Criteria Not Met | 0
  Artery and Vein: STAGE R2*MAP Criteria Met | 89
  Artery and Vein: STAGE R2*MAP Criteria Not Met | 0
  Artery and Vein: STAGE T2*MAP Criteria Met | 89
  Artery and Vein: STAGE T2*MAP Criteria Not Met | 0
  Artery and Vein: STAGE MRA Criteria Met | 89
  Artery and Vein: STAGE MRA Criteria Not Met | 0
  Artery and Vein: STAGE pSWIM Criteria Met | 89
  Artery and Vein: STAGE pSWIM Criteria Not Met | 0
  Artery and Vein: STAGE mpSWIM Criteria Met | 89
  Artery and Vein: STAGE mpSWIM Criteria Not Met | 0
  Artery and Vein: STAGE T1WE Criteria Met | NA — T1WE can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE T1WE Criteria Not Met | NA — T1WE can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE T1MAP Criteria Met | NA — T1MAP can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE T1MAP Criteria Not Met | NA — T1MAP can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE PDMAP Criteria Met | NA — PDMAP can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE PDMAP Criteria Not Met | NA — PDMAP can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE DIR Criteria Met | NA — DIR can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Artery and Vein: STAGE DIR Criteria Not Met | NA — DIR can not be properly assessed for Artery/Vein appearance due to the lack of signal in Artery/Vein in the image series.
  Calcium and Iron: Conventional T1MPRAGE Criteria Met | 89
  Calcium and Iron: Conventional T1MPRAGE Criteria Not Met | 0
  Calcium and Iron: Conventional T1W Criteria Met | 89
  Calcium and Iron: Conventional T1W Criteria Not Met | 0
  Calcium and Iron: Conventional PDW Criteria Met | 89
  Calcium and Iron: Conventional PDW Criteria Not Met | 0
  Calcium and Iron: STAGE T1W Criteria Met | 89
  Calcium and Iron: STAGE T1W Criteria Not Met | 0
  Calcium and Iron: STAGE PDW Criteria Met | 89
  Calcium and Iron: STAGE PDW Criteria Not Met | 0
  Calcium and Iron: STAGE SWI Criteria Met | 89
  Calcium and Iron: STAGE SWI Criteria Not Met | 0
  Calcium and Iron: STAGE tSWI Criteria Met | 89
  Calcium and Iron: STAGE tSWI Criteria Not Met | 0
  Calcium and Iron: STAGE iSWIM Criteria Met | 89
  Calcium and Iron: STAGE iSWIM Criteria Not Met | 0
  Calcium and Iron: STAGE R2*MAP Criteria Met | 89
  Calcium and Iron: STAGE R2*MAP Criteria Not Met | 0
  Calcium and Iron: STAGE T2*MAP Criteria Met | 89
  Calcium and Iron: STAGE T2*MAP Criteria Not Met | 0
  Calcium and Iron: STAGE MRA Criteria Met | NA — MRA can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE MRA Criteria Not Met | NA — MRA can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE pSWIM Criteria Met | 89
  Calcium and Iron: STAGE pSWIM Criteria Not Met | 0
  Calcium and Iron: STAGE mpSWIM Criteria Met | 89
  Calcium and Iron: STAGE mpSWIM Criteria Not Met | 0
  Calcium and Iron: STAGE T1WE Criteria Met | NA — T1WE can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE T1WE Criteria Not Met | NA — T1WE can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE T1MAP Criteria Met | NA — T1MAP can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE T1MAP Criteria Not Met | NA — T1MAP can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE PDMAP Criteria Met | NA — PDMAP can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE PDMAP Criteria Not Met | NA — PDMAP can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE DIR Criteria Met | NA — DIR can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Calcium and Iron: STAGE DIR Criteria Not Met | NA — DIR can not be properly assessed for Calcium/Iron appearance due to the lack of signal from Calcium/Iron in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: Conventional T1MPRAGE Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: Conventional T1MPRAGE Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: Conventional T1W Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: Conventional T1W Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: Conventional PDW Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: Conventional PDW Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T1W Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T1W Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE PDW Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE PDW Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE SWI Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE SWI Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE tSWI Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE tSWI Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE iSWIM Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE iSWIM Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE R2*MAP Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE R2*MAP Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T2*MAP Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T2*MAP Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE MRA Criteria Met | NA — MRA can not be properly assessed for GM/WM/CSF appearance due to the lack of signal from GM/WM/CSF contrast in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE MRA Criteria Not Met | NA — MRA can not be properly assessed for GM/WM/CSF appearance due to the lack of signal from GM/WM/CSF contrast in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE pSWIM Criteria Met | NA — pSWIM can not be properly assessed for GM/WM/CSF appearance due to the lack of signal from GM/WM/CSF contrast in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE pSWIM Criteria Not Met | NA — pSWIM can not be properly assessed for GM/WM/CSF appearance due to the lack of signal from GM/WM/CSF contrast in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE mpSWIM Criteria Met | NA — mpSWIM can not be properly assessed for GM/WM/CSF appearance due to the lack of signal from GM/WM/CSF contrast in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE mpSWIM Criteria Not Met | NA — mpSWIM can not be properly assessed for GM/WM/CSF appearance due to the lack of signal from GM/WM/CSF contrast in the image series.
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T1WE Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T1WE Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T1MAP Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE T1MAP Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE PDMAP Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE PDMAP Criteria Not Met | 0
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE DIR Criteria Met | 89
  Gray Matter / White Matter / Cerebrospinal Fluid: STAGE DIR Criteria Not Met | 0

4. Primary Outcome: Evaluation of STAGE Image Processing Times
Description: Review of the recorded processing times for the STAGE module to accept and process STAGE inputs and to export them back to the PACS as STAGE outputs.
Time Frame: Baseline Only
Population: The average and minimum/maximum processing times for STAGE were evaluated across scanners, resolutions, and field strengths.
Measure: Mean (Standard Deviation); unit: Time (minutes)
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
Number analyzed (Participants) | 89
Time (minutes)
  3T GE Signa Premier: number analyzed (Participants) | 44
  3T GE Signa Premier | 17.4 (3.2)
  1.5T Siemens Aera: number analyzed (Participants) | 20
  1.5T Siemens Aera | 7.6 (0.8)
  3T Siemens Skyra: number analyzed (Participants) | 20
  3T Siemens Skyra | 10.1 (1.7)
  3T Siemens Prisma: number analyzed (Participants) | 5
  3T Siemens Prisma | 11.3 (2.0)

ADVERSE EVENTS:
Time Frame: Adverse event data collected per MRI routine examination, approximately up to 90 minutes. Participants were observed during the MRI scan. No follow-up data were recorded.
Arm/Group | STrategically Acquired Gradient Echo (STAGE)
All-Cause Mortality (participants affected / at risk) | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92
Other Adverse Events (participants affected / at risk) | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-10): https://cdn.clinicaltrials.gov/large-docs/01/NCT04292301/Prot_SAP_002.pdf
  • Informed Consent Form (2020-01-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT04292301/ICF_001.pdf